CLINICAL TRIAL: NCT06586320
Title: Using Mathematical Quantification of Limb and Eye Movements of Parkinson's Disease Patients As a Biomarker for Classification and Prediction of Disease State and Response to Treatment
Brief Title: Quantification of Parkinson's Disease Patients As a Biomarker for Classification, Prediction and Response to Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stardots AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUS-001; STUDY02002335 (Other: Dartmouth-Hitchcock)
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Quantification; Biomarker; Classification
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- ON, One visit (Other): Subject visit one time at clinic for tests and assessments. Subject type are Essential Tremor (ET), Healthy Control (HC) or Idiopathic Parkinson's Disease (IPD).
  The first arm will include the majority of subjects that will be enrolled in a onetime only study procedure performance. Subjects of this arm will carry the diagnosis of IPD, ET, or HC. After the completion of their first research visit and completing study procedures, there will be no future visits or procedures.
  Interventions: Device: Evaluation of mathematical models
- OFF/ON (Other): Subject visit one time at clinic for tests and assessments without medication, carry out tests and assessments, then take medication according to the protocol, then carry our tests and assessments.
  Subject type are Idiopathic Parkinson's Disease.
  Interventions: Drug: 150% of their routine home dopaminergic medications dose right in the clinic; Device: Evaluation of mathematical models
- ON, Longitudinal (Other): IPD subjects will be asked to repeat the study visit and procedures every 6 months for longitudinal monitoring.
  Interventions: Device: Evaluation of mathematical models

INTERVENTIONS:
Drug: 150% of their routine home dopaminergic medications dose right in the clinic — IPD subjects will be informed head of time not to take their dopaminergic medications and other Parkinson's non-dopaminergic medications such as anticholinergics, NMDA inhibitors, and adenosine blockers for at least 12 hours prior to their initial procedure. Immediately, after conducting both hand movement and eye movement tests, the patient will take 150% of their routine home dopaminergic medications dose right in the clinic. They will also take their non-dopaminergic medications doses similar to home dose with no change. This will be under the supervision of their treating movement disorders specialist and study PI.
  Arms: OFF/ON
Device: Evaluation of mathematical models — Evaluation of performance of mathematical models developed to quantify and classify symptoms and disease state using sensor data from smart phone and eye tracking cameras

SUMMARY:
This is a three-armed open investigational study that aims to differentiate, quantify, and categorize abnormal eye movements and upper limbs movements in patients with Parkinson's disease. The study is using investigational non-invasive devices for that reason including ANLIVA® Hand Movement and ANLIVA® Eye Movement.

DETAILED DESCRIPTION:
To evaluate performance of mathematical models developed to quantify and classify symptoms and disease state using sensor data from smart phone and eye tracking cameras in subjects with Parkinson's disease.

A clinical investigator will be capturing data from the clinical encounter completed by default the same day in addition to other clinical questionnaires subjects will be filling themselves. A percentage of subjects will be asked prior to their arrival to be part of a subset study called OFF/ON study, where they will be asked not to take their IPD oral home medications prior to arrival. Both study procedure elements will be performed at the beginning of the evaluation and 60 minutes after taking their medication. There is also a longitudinal study part, where a percentage of the subjects will be asked to visit the clinic with 6 months interval, up to 4 times, including the first visit. There will be a percentage of approached subjects that belong to the category of Essential Tremor (ET) and Healthy control (HC) used for comparison purposes. ET and HC subjects will undergo the same recruitment and testing process.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the investigation, the subjects must fulfil all the below criteria prior to enrolment:

1. Subjects already diagnosed with Idiopathic Parkinson's Disease (IPD)
2. or subjects already diagnosed with Essential tremor (ET)
3. or subjects who are healthy controls (HC) and are not diagnosed with IPD or ET
4. Able to understand and sign the informed consent form.

Exclusion Criteria:

Subjects that meet any of the below criteria will be excluded:

1. Not able to sign the informed consent form
2. Below 18 years of age
3. Diagnosed with movement disorder other than IPD or ET that might interfere with hand movements or eye movements (tics, myoclonus, chorea, dystonia, etc)
4. Has parkinsonism not due to IPD (drug induced, functional, vascular, etc)
5. Visual or physical limitations that prevent the subject from performing the baseline eye study requirements
6. Being involved in the planning and conduct of the clinical investigation (applies to all sponsor management staff, investigational staff and third-party vendors as applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of current IPD motor symptoms using kinetic tremor and Dyskinesia test | Day 1
  ANLIVA® Hand Movement score of kinetic tremor test and dyskinesia test will be measured. Measurements are done on subjects upper limb movements. SD score of kinetic tremor test and dyskinesia test will be assessed by assessors.
  SD is acronym for Stardots-Dartmouth score. The SD score will be used to benchmark the ANLIVA® device assessments as a nonreference standard.
  Minimum value is 0; maximum value is 4. A higher value on the SD score means more movement disorder.

SECONDARY OUTCOMES:
Quantification of current IPD motor symptoms using rest tremor and postural tremor test | Day 1
  ANLIVA® Hand Movement score of rest tremor test and postural test will be measured. Measurements are done on subjects upper limb movements. SD score of rest test and postural tremor test will be assessed by assessors.
  SD is acronym for Stardots-Dartmouth score. The SD score will be used to benchmark the ANLIVA® device assessments as a nonreference standard.
  Minimum value is 0; maximum value is 4. A higher value on the SD score means more movement disorder.
Classification between Dyskinesia or kinetic tremor | Day 1
  ANLIVA® Hand Movement score of kinetic tremor test and dyskinesia test will be measured. Measurements are done on subjects upper limb movements. This will be compared to assessments of SD score Dyskinesia classification.
  SD is acronym for Stardots-Dartmouth score. The SD score will be used to benchmark the ANLIVA® device assessments as a nonreference standard.
  Minimum value is 0; maximum value is 4. A higher value on the SD score means more movement disorder.

OTHER OUTCOMES:
Collect data for developing test for bradykinesia (exploratory) | Day 1
  Bradykinesia part of ANLIVA® Hand Movement will be measured. Measurements are done on subjects upper limb movements.
Derive optimized variables for objective quantification and/or classification of ocular movements (exploratory) | Day 1
  Ocular movements will be measured using ANLIVA® Eye Movement. Measurements are done on subjects eye movements

CONTACTS AND LOCATIONS:
Overall Officials: Anas Hannoun, MD, Principal Investigator — Dartmouth Hitchcock medical center, Manchester
Locations (1):
- Dartmouth Hitchcock medical center, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No